CLINICAL TRIAL: NCT01451411
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled, Multi-Center, Dose-Titration Study to Assess the Efficacy, Safety and Pharmacokinetics of Intravenous Conivaptan (Vaprisol®) in Pediatric Subjects With Euvolemic or Hypervolemic Hyponatremia
Brief Title: A Study to Assess the Efficacy, Safety and Pharmacokinetics of Intravenous Conivaptan (Vaprisol®) in Pediatric Subjects With Euvolemic or Hypervolemic Hyponatremia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment goals were not met.
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 087-CL-096
Record Dates: First submitted 2011-10-05; First posted 2011-10-13 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Hyponatremia
Keywords: Serum Sodium; Euvolemia; Hypervolemia; Vaprisol®; Conivaptan; YM087
MeSH Terms: conditions — Hyponatremia; Edema | interventions — conivaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conivaptan hydrochloride (Experimental)
  Interventions: Drug: Conivaptan hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Conivaptan hydrochloride — Intravenous
  Other Names: Vaprisol®; YM087
  Arms: Conivaptan hydrochloride
Drug: Placebo — Intravenous
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy, safety and pharmacokinetics of intravenous conivaptan in pediatric subjects with abnormally low concentration of sodium in blood.

DETAILED DESCRIPTION:
A 3:1 randomization between conivaptan and placebo will be implemented and randomization will be further stratified in a 1:1:2 ratio for age groups: 2-5 years, 6-10 years, and 11-17 years.

Subjects will need to remain hospitalized for the 48-hour Treatment Period through Hour 96 (Day 4). There will be a follow-up safety visit on Day 9 or day of hospital discharge, whichever occurs first. There is a final follow-up phone call at Day 32 to assess if any serious adverse events have occurred since hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Subject is euvolemic or hypervolemic hyponatremia upon clinical presentation
* Subject has serum sodium value ≥ 115 mEq/L (115 mmol/L) and < 130 mEq/L (130 mmol/L) during the 24 hours preceding inclusion into the study
* Female subject of childbearing potential must have a negative serum pregnancy test and must be premenarchal, surgically sterile or must practice a method of birth control

Exclusion Criteria:

* Female subject is pregnant or lactating
* Subject has a body mass index (BMI) < the 3rd percentile or > the 97th percentile for their age and stature according to the World Health Organization; Body mass index-for-age percentiles charts for boys and girls ages 2 to 20
* Subject has clinical evidence of volume depletion, dehydration or hypovolemia
* Subject with hypovolemic hyponatremia or transient causes of hyponatremia that are likely to resolve during the time of study participation
* Subjects with a cause of hyponatremia that is most appropriately corrected by alternative therapies
* Subject is expected to receive emergent treatment for hyponatremia during the treatment period of the study
* Subject has clinical evidence of hypotension
* Subject has uncontrolled hypertension > the 99th percentile for their age
* Subject has uncontrolled bradyarrhythmias or tachyarrhythmias requiring emergent pacemaker placement or treatment
* Subject has untreated severe hypothyroidism, hyperthyroidism or adrenal insufficiency
* Subject has known urinary outflow obstruction, unless subject is, or can be catheterized during the study
* Subject has estimated creatinine clearance < 30 mL/min during the seven days prior to study drug administration
* Subject has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevations > 3 times the upper limit of normal reference range during the seven days prior to study drug administration
* Subject has serum albumin ≤ 1.5 g/dL during the seven days prior to study drug administration
* Subject has white blood cell count (WBC) < 3000/micro-liter documented any time during seven days prior to study drug administration or anticipated drop in WBC to < 3000/micro-liter during the period of the study due to chemotherapy
* Subject currently has unstable hepatic function or a history of hepatic encephalopathy, or bleeding esophageal varices within the last 3 months
* Subject has acute heart failure. Prior history of heart failure is allowed if there are no current signs/symptoms
* Subject has a non-fasting blood glucose value ≥ 275 mg/dL
* Subject requires or is suspected to require treatment with potent inhibitors or potent inducers of CYP3A4
* Subject was administered hypertonic saline or oral salt supplement within 24 hours prior to study drug administration
* Subject requires the use of medications used in the treatment of Syndrome of Inappropriate Antidiuretic Hormone Secretion (SIADH): including lithium salts, urea or demeclocycline during the week prior to screening and throughout the study drug treatment period
* Subject has any condition that may interfere with treatment or evaluation of safety
* Subject has received investigational therapy (including placebo) within 28 days or 5 half lives, whichever is longer

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (3):
- Children's Hospital of New York - Presbyterian, New York, New York, United States
- Colombia (2):
  - Fundación Cardioinfantil - Instituto Cardiológico, Bogotá
  - Fundación Valle del Lili, Cali, Valle

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conivaptan Hydrochloride | Placebo
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conivaptan Hydrochloride | Placebo | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Customized [Number; unit: participants]
  2 - 5 years | 0 | 0 | 0
  6 - 10 years | 2 | 0 | 2
  11 - 17 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Colombia | 2 | 0 | 2
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to the End of the 48-hour Treatment Period in Serum Sodium
Time Frame: baseline and 48 hours
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Conivaptan Hydrochloride | Placebo
Number analyzed (Participants) | 3 | 1
mEq/L | 6.0 (5.3) | -4.0

2. Secondary Outcome: Time From the First Dose of Study Medication to a Confirmed ≥ 4 mEq/L Increase From Baseline in Serum Sodium
Time Frame: 48 hours
Population: Data from two subjects (one conivaptan, and one placebo) were censored as the serum sodium never achieved a value greater or equal to 4 mEq/L above the baseline value.
Measure: Mean (Full Range); unit: hours
Arm/Group | Conivaptan Hydrochloride | Placebo
Number analyzed (Participants) | 2 | 0
hours | 21.5 [2.5 to 40.5] |

3. Secondary Outcome: Number of Patients With Confirmed ≥ 4 mEq/L Increase From Baseline in Serum Sodium
Time Frame: baseline and 48 hours
Measure: Number; unit: participants
Arm/Group | Conivaptan Hydrochloride | Placebo
Number analyzed (Participants) | 3 | 1
participants | 2 | 0

4. Secondary Outcome: Number of Subjects With Confirmed > 6 mEq/L Increase From Baseline in Serum Sodium or a Confirmed Normal Serum Sodium Level (Greater Than or Equal to 135 mEq/L)
Time Frame: baseline and 48 hours
Measure: Number; unit: participants
Arm/Group | Conivaptan Hydrochloride | Placebo
Number analyzed (Participants) | 3 | 1
participants | 1 | 0

5. Secondary Outcome: Change From Baseline in Effective Water Clearance (EWC) Every 12 Hours
Time Frame: Baseline, Hours 12, 24, 36 and 48
Population: The protocol specifies that calculations for this endpoint were to be derived by the statistical team. Due to the terminated status of the study, a statistical team was not employed and calculations to determine this variable were not performed.
Arm/Group | Conivaptan Hydrochloride | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Free Water Clearance (FWC)
Time Frame: Baseline and 48 hours
Population: as for outcome 5
Arm/Group | Conivaptan Hydrochloride | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With an Overly Rapid Rise in Serum Sodium From Baseline
Description: an absolute serum sodium of 145 mEq/L at Hour 24 or an increase in serum sodium of greater than 12 mEq/L
Time Frame: baseline and Hours 3, 8, 12 and 24.
Measure: Number; unit: participants
Arm/Group | Conivaptan Hydrochloride | Placebo
Number analyzed (Participants) | 3 | 1
participants | 0 | 0

8. Secondary Outcome: Population Pharmacokinetics: Clearance (CL)
Description: Based on conivaptan concentrations, the pharmacokinetics of the study population will be analyzed to determine median CL
Time Frame: Up to Hour 60
Population: Due to the terminated status of the study, pharmacokinetic samples were not analyzed.
Arm/Group | Conivaptan Hydrochloride | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Population Pharmacokinetics: Volume of Distribution (Vd)
Description: Based on conivaptan concentrations, the pharmacokinetics of the study population will be analyzed to determine median Vd
Time Frame: Up to Hour 60
Population: Due to the terminated status of the study, pharmacokinetic samples were not analyzed.
Arm/Group | Conivaptan Hydrochloride | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Through Day 32
Description: Serious adverse events were collected through Day 32; non-serious adverse events were collected through Day 9.
Arm/Group | Conivaptan Hydrochloride | Placebo
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 2/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conivaptan Hydrochloride (N=3) | Placebo (N=1)
Stevens_Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Onset of SAE was on Day 32 following initiation of investigational drug. The event was deemed as not related by the Investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conivaptan Hydrochloride (N=3) | Placebo (N=1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Accelerated idioventricular rhythm (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish data generated at their study site after multi-center study data have already been published, or after 18 months have elapsed following database lock, whichever comes first. The sponsor may review manuscripts before submission and delay publication by an additional 60 days, if necessary.